CLINICAL TRIAL: NCT01904149
Title: A Randomized, Double-blind, Placebo and Active-controlled, Parallel-group Study to Evaluate the Analgesic Efficacy and Safety of Dexketoprofen Trometamol and Tramadol Hydrochloride Oral Fixed Combination on Moderate to Severe Acute Pain Following Abdominal Hysterectomy
Brief Title: Oral Treatment for Gynaecological Post-operative Pain With Dexketoprofen Trometamol and Tramadol Hydrochloride
Acronym: DAVID lap
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEX-TRA-04; 2012-004545-32 (EudraCT Number)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Acute Pain
Keywords: Moderate to severe acute pain; Postoperative pain; Abdominal hysterectomy; Analgesics; Dexketoprofen; Tramadol
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- DKP/TRAM followed by DKP/TRAM (Experimental): Dexketoprofen/Tramadol-single dose followed by Dexketoprofen/Tramadol-multiple doses
  Interventions: Drug: Dexketoprofen/Tramadol-single dose; Drug: Dexketoprofen/Tramadol-multiple doses
- DKP followed by DKP (Active Comparator): Dexketoprofen-single dose followed by Dexketoprofen-multiple doses
  Interventions: Drug: Dexketoprofen-single dose; Drug: Dexketoprofen-multiple doses
- TRAM followed by TRAM (Active Comparator): Tramadol-single dose followed by Tramadol-multiple doses
  Interventions: Drug: Tramadol-single dose; Drug: Tramadol-multiple doses
- Placebo followed by DKP/TRAM (Other): Placebo single dose followed by Dexketoprofen/Tramadol-multiple doses
  Interventions: Drug: Placebo; Drug: Dexketoprofen/Tramadol-multiple doses
- Placebo followed by DKP (Other): Placebo single dose followed by Dexketoprofen-multiple doses
  Interventions: Drug: Placebo; Drug: Dexketoprofen-multiple doses
- Placebo followed by TRAM (Other): Placebo single dose followed by Tramadol-multiple doses
  Interventions: Drug: Placebo; Drug: Tramadol-multiple doses

INTERVENTIONS:
Drug: Placebo — Placebo single oral dose (first 8 hours)
  Arms: Placebo followed by DKP; Placebo followed by DKP/TRAM; Placebo followed by TRAM
Drug: Dexketoprofen-single dose — Dexketoprofen single oral dose (first 8 hours)
  Arms: DKP followed by DKP
Drug: Tramadol-single dose — Tramadol single oral dose (first 8 hours)
  Arms: TRAM followed by TRAM
Drug: Dexketoprofen/Tramadol-single dose — Dexketoprofen/Tramadol single oral dose (first 8 hours)
  Arms: DKP/TRAM followed by DKP/TRAM
Drug: Dexketoprofen-multiple doses — Dexketoprofen multiple oral doses t.i.d. for 3 days (total 6 doses)
  Arms: DKP followed by DKP; Placebo followed by DKP
Drug: Tramadol-multiple doses — Tramadol multiple oral doses t.i.d. for 3 days (total 6 doses)
  Arms: Placebo followed by TRAM; TRAM followed by TRAM
Drug: Dexketoprofen/Tramadol-multiple doses — Dexketoprofen/Tramadol multiple oral doses t.i.d. for 3 days (total 6 doses)
  Arms: DKP/TRAM followed by DKP/TRAM; Placebo followed by DKP/TRAM

SUMMARY:
This study aims to evaluate the analgesic efficacy of single and repeated doses of fixed combination of dexketoprofen trometamol (DKP) and tramadol hydrochloride (TRAM) in comparison to the single agents (and placebo for the single dose phase only).

Approximately 600 female patients presenting moderate to severe pain after a total/subtotal abdominal hysterectomy are eligible to be randomised provided that they experience moderate to severe pain on the day after surgery.

DETAILED DESCRIPTION:
In this clinical trial patients were randomized to the described 6 treatment arms, where each arm define the treatment to be received in the first single dose phase (lasting 8 hours after the 1st treatment intake) and in the subsequent multiple-dose phase (lasting from the second treatment intake up to the 8 hours after the last intake). Namely:

* DKP/TRAM followed by DKP/TRAM;
* DKP followed by DKP;
* TRAM followed by TRAM;
* placebo followed by DKP;
* placebo followed by TRAM;
* placebo followed by DKP/TRAM;

The analyses of endpoints pertinent to the single dose phase were performed combining all the 3 treatment arms including placebo into one group, which resulted in the following 4 analysis groups: DKP/TRAM, DEXKETOPROFEN, TRAMADOL, and Placebo.

The analysis of endpoints pertinent to the multiple dose phase were performed combining the treatment arms including the same active treatment, which resulted in the following 3 analysis groups: DKP/TRAM, DEXKETOPROFEN, and TRAMADOL.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 75 years.
* Scheduled to undergo a total or subtotal abdominal hysterectomy (with or without salpingo-oophorectomy) for benign conditions.
* Patients experiencing pain at rest of at least moderate intensity the day after surgery.

Exclusion Criteria:

* Patients not suitable for study treatments and rescue medication (RM) or those for whom non-steroidal anti-inflammatory drugs (NSAIDs), opioids, acetyl salicylic acid, pyrazolones or pyrazolidines are contraindicated.
* Patients with clinically significant abnormalities in vital signs, safety laboratory tests and 12-lead ECG at screening.
* Patients with history of any illness or condition that might pose a risk to the patient or confound the efficacy and safety study results.
* Patients using and not suitable to withdraw analgesics other than those specified in the protocol.
* Patients using and not suitable for withdrawing any of the prohibited medication specified in the protocol.
* Breastfeeding women.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry J McQuay, Professor, Study Chair — Balliol College Oxford; Andrew Moore, Professor, Study Chair — Pain Research & Nuffield Department of Anaesthetics - University of Oxford
Locations (28):
- Hungary (4):
  - Bajcsy-Zsilinszky Kórház, Budapest
  - University Hospital of Debrecen, Debrecen
  - Dr. Bugyi István Kórház, Szentes
  - Fejér megyei Szent György Kórház, Székesfehérvár
- Latvia (2):
  - Juras Medicinas Centre, Riga
  - Riga East University Hospital Gynecology Clinic, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Vilniaus gimdymo namai, Vilnius
- Poland (8):
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Prywatna Klinika Polozniczo-Ginekologiczna, Bialystok
  - Ginekologiczno-Polożniczy Szpital Kliniczny UM w Poznaniu, Poznan
  - Wojewodzki Szpital, Przemyśl
  - Specjalistyczny Szpital im. E. Szczeklika, Tarnów
  - Wojskowy Instytut Medyczny, Centralny Szpital Kliniczny Mini, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
- Romania (7):
  - Institutul pentru Ocrotirea Mamei si Copilului (IOMC) "Prof. Dr. Alfred Rusescu", Bucharest
  - Genesys Fertility Center, Bucharest
  - Spitalul Clinic "Dr. Ioan Cantacuzino" - Sectia Clinica Obstetrica Ginecologie II, Bucharest
  - Spitalul Clinic "Dr. Ioan Cantacuzino" - Sectia Clinica Obstetrica Ginecologie I, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic de Urgenta "Sfantul Pantelimon", Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures - Sectia Obstretica Ginecologie I, Târgu Mureş
- Russia (2):
  - Moscow Regional Research Institute of Obstetrics and Gynecol, Moscow
  - FGUZ Clinical Hospital 122 n.a. L.G. Sokolova FMBA, Saint Petersburg
- GYNPOR, s.r.o., Sliač, Slovakia
- Spain (2):
  - Hospital Universitario Arnau de Vilanova, Lleida, Lérida
  - Complejo Hospitalario Arquitecto Marcide, Ferrol

REFERENCES:
- [Result] Moore RA, McQuay HJ, Tomaszewski J, Raba G, Tutunaru D, Lietuviete N, Galad J, Hagymasy L, Melka D, Kotarski J, Rechberger T, Fulesdi B, Nizzardo A, Guerrero-Bayon C, Cuadripani S, Piza-Vallespir B, Bertolotti M. Dexketoprofen/tramadol 25 mg/75 mg: randomised double-blind trial in moderate-to-severe acute pain after abdominal hysterectomy. BMC Anesthesiol. 2016 Jan 22;16:9. doi: 10.1186/s12871-016-0174-5. PMID 26801905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DKP/TRAM Followed by DKP/TRAM | DKP Followed by DKP | TRAM Followed by TRAM | Placebo Followed by DKP/TRAM | Placebo Followed by DKP | Placebo Followed by TRAM
Started | 152 | 151 | 150 | 51 | 51 | 51
Single-dose Phase | 152 | 151 | 150 | 51 | 51 | 51
Multiple-dose Phase | 150 | 146 | 149 | 48 | 48 | 49
Completed | 147 | 140 | 148 | 47 | 46 | 48
Not Completed | 5 | 11 | 2 | 4 | 5 | 3
Not completed — Adverse Event | 3 | 4 | 0 | 1 | 1 | 2
Not completed — Lack of Efficacy | 0 | 3 | 1 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — non compliance with study drug | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population (which includes all patients randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | DKP/TRAM Followed by DKP/TRAM | DKP Followed by DKP | TRAM Followed by TRAM | Placebo Followed by DKP/TRAM | Placebo Followed by DKP | Placebo Followed by TRAM | Total
Number analyzed (Participants) | 152 | 151 | 150 | 51 | 51 | 51 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (6.70) | 47.2 (7.07) | 47.6 (6.87) | 47.4 (6.82) | 47.4 (7.46) | 47.2 (4.60) | 47.6 (6.75)
Sex/Gender, Customized [Number; unit: participants]
  Females | 152 | 151 | 150 | 51 | 51 | 51 | 606
Race/Ethnicity, Customized [Number; unit: participants]
  White | 152 | 151 | 150 | 51 | 51 | 51 | 606
Region of Enrollment [Number; unit: participants]
  Hungary | 22 | 19 | 26 | 8 | 7 | 7 | 89
  Slovakia | 7 | 13 | 8 | 5 | 2 | 4 | 39
  Spain | 1 | 2 | 1 | 0 | 0 | 1 | 5
  Poland | 63 | 53 | 60 | 18 | 23 | 17 | 234
  Romania | 32 | 40 | 32 | 10 | 12 | 12 | 138
  Lithuania | 2 | 4 | 3 | 1 | 1 | 3 | 14
  Russian Federation | 3 | 3 | 3 | 2 | 2 | 2 | 15
  Latvia | 22 | 17 | 17 | 7 | 4 | 5 | 72
Weight [Mean (Standard Deviation); unit: kg] | 75.2 (15.15) | 72.1 (13.54) | 71.3 (12.17) | 73.6 (13.74) | 72.9 (14.60) | 72.6 (10.97) | 72.9 (13.58)
Height [Mean (Standard Deviation); unit: cm] | 163.9 (5.40) | 163.7 (6.37) | 164.1 (6.10) | 164.5 (6.17) | 163.5 (5.94) | 164.4 (5.59) | 164.0 (5.94)

OUTCOME MEASURES:

1. Primary Outcome: SPID8 (Sum of Pain Intensity Differences Over 8 Hours)
Description: Sum of Pain Intensity Differences calculated as the weighted sum of the PI-VAS differences over 8 hour period. PI-VAS corresponds to the pain intensity measured by a 0-100 visual analogue scale (0=no pain to 100=worst pain imaginable) which was measured at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, and 8h after the first dose. A higher value in SPID indicates greater pain relief.
  The analysis was performed combining all randomization arms including placebo into one group, which resulted in the following 4 analysis groups: DKP/TRAM, DEXKETOPROFEN, TRAMADOL, and Placebo.
Time Frame: over 8 hours after the first dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DKP/TRAM: Drug: Dexketoprofen/Tramadol single oral dose (first 8 hours) Arm type: experimental; Dexketoprofen/Tramadol single oral dose (first 8 hours)
- DEXKETOPROFEN: Drug: Dexketoprofen single oral dose (first 8 hours) Arm type: active comparator; Dexketoprofen single oral dose (first 8 hours)
- TRAMADOL: Drug: Tramadol single oral dose (first 8 hours) Arm type: active comparator; Tramadol single oral dose (first 8 hours)
- PLACEBO: Drug: Placebo single oral dose (first 8 hours) Arm type: Placebo comparator; Placebo single oral dose (first 8 hours)
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL | PLACEBO
Number analyzed (Participants) | 152 | 151 | 150 | 153
units on a scale | 241.8 (139.06) | 184.5 (139.23) | 157.3 (150.89) | 117.0 (121.80)

2. Secondary Outcome: Percentage of Responders According to 50% Max TOTPAR (Total Pain Relief)
Description: Percentage of responders over 8 hours after first dose, according to the 50% maximum total pain relief rule: maximum TOTPAR calculated as the theoretical maximum weighted sum of PAR-VRS (Pain Relief - Verbal Rating Scale: pain relief 0=none, 4=complete) scores.
  The analysis was performed combining all randomization arms including placebo into one group, which resulted in the following 4 analysis groups: DKP/TRAM, DEXKETOPROFEN, TRAMADOL, and Placebo.
Time Frame: over 8 hours after first dose
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- PLACEBO: Drug: Placebo; Arm type: PLACEBO comparator; Placebo single oral dose during single dose phase (first 8 hours); Drug: Placebo single oral dose (first 8 hours) Arm type: placebo comparator; placebo single oral dose (first 8 hours)
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL | PLACEBO
Number analyzed (Participants) | 152 | 151 | 150 | 153
percentage of participants | 65.8 | 47.7 | 44.0 | 30.7

3. Secondary Outcome: SPID48 (Sum of Pain Intensity Differences Over 48 Hours of the Multiple-dose Phase)
Description: Sum of Pain Intensity Differences calculated as the weighted sum of the PI-VAS differences over 48 hours of the multiple-dose phase.
  PI-VAS corresponds to the pain intensity measured by a 0-100 visual analogue scale (0=no pain to 100=worst pain imaginable) which was measured every two hours over the first 48 hours of the multiple-dose phase. A higher value in SPID indicates greater pain relief.
  The analysis was performed combining all randomization arms including the same active treatment, which resulted in the following 3 analysis groups: DKP/TRAM, DEXKETOPROFEN, and TRAMADOL.
Time Frame: over 48 hours of the multiple-dose phase
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DKP/TRAM: Drug: Dexketoprofen/Tramadol multiple doses; Arm type: experimental; Dexketoprofen/Tramadol multiple oral doses t.i.d. for 3 days (a total of 6 doses)
- DEXKETOPROFEN: Drug: Dexketoprofen multiple doses; Arm type: active comparator; Dexketoprofen multiple oral doses t.i.d. for 3 days (a total of 6 doses)
- TRAMADOL: Drug: Tramadol multiple doses; Arm type: active comparator; Tramadol multiple oral doses t.i.d. for 3 days (a total of 6 doses)
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL
Number analyzed (Participants) | 203 | 202 | 201
units on a scale | 2273.0 (864.03) | 1965.2 (912.19) | 2035.0 (919.49)

4. Secondary Outcome: Percentage of Responders According to PI-VAS (Pain Intensity - Visual Analogue Scale)
Description: Percentage of responders; response defined as achievement a mean pain intensity, PI-VAS < 40 mm (PI-VAS corresponds to the pain intensity measured by a 0-100 visual analogue scale, 0=no pain to 100=worst pain imaginable), over 48 hours of the multiple-dose phase.
  The analysis was performed combining all randomization arms including the same active treatment, which resulted in the following 3 analysis groups: DKP/TRAM, DEXKETOPROFEN, and TRAMADOL.
Time Frame: over 48 hours of the multiple-dose phase
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | DKP/TRAM | DEXKETOPROFEN | TRAMADOL
Number analyzed (Participants) | 203 | 202 | 201
percentage of participants | 94.1 | 82.7 | 88.6

ADVERSE EVENTS:
Time Frame: Study duration for patients was up to 6 weeks
Description: Analyzed for the Safety population (all patients randomized who received at least one dose of the study treatment). Includes adverse events emerging after at least one dose of active study treatment.
Arm/Group | DKP/TRAM Followed by DKP/TRAM | DKP Followed by DKP | TRAM Followed by TRAM | Placebo Followed by DKP/TRAM | Placebo Followed by DKP | Placebo Followed by TRAM
Serious Adverse Events (participants affected / at risk) | 7/151 | 2/152 | 1/150 | 0/52 | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 22/151 | 22/152 | 33/150 | 3/52 | 10/50 | 10/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DKP/TRAM Followed by DKP/TRAM (N=151) | DKP Followed by DKP (N=152) | TRAM Followed by TRAM (N=150) | Placebo Followed by DKP/TRAM (N=52) | Placebo Followed by DKP (N=50) | Placebo Followed by TRAM (N=51)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscense (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
peritoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fallopian tube torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laparotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer stage I (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The investigator assessed the event as non serious. However, the event seriousness was upgraded by the sponsor as "other medically important condition".
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DKP/TRAM Followed by DKP/TRAM (N=151) | DKP Followed by DKP (N=152) | TRAM Followed by TRAM (N=150) | Placebo Followed by DKP/TRAM (N=52) | Placebo Followed by DKP (N=50) | Placebo Followed by TRAM (N=51)
Nausea (Gastrointestinal disorders) | 9 (10) | 6 (7) | 14 (15) | 3 (3) | 2 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (6) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2) | 6 (6) | 0 (0) | 2 (2) | 3 (3)
Platelet count increased (Investigations) | 3 (3) | 8 (8) | 9 (9) | 0 (0) | 3 (3) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the PI will allow the Sponsor at least 60 days to review and comment upon the publication manuscript. The Sponsor will provide any manuscript of the results of this study at least 60 days before publishing to the authors for a complete review.